CLINICAL TRIAL: NCT02407483
Title: Laparoscopic Simulator Training With or Without Laser Visual Guidance -A Randomized Trial
Brief Title: Laparoscopic Training With Laser Guidance Trial
Acronym: LVG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Stine Maya Dreier Sørensen, Medical Student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014-6022
Record Dates: First submitted 2015-03-19; First posted 2015-04-03 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Depth Perception
Keywords: Laparoscopy; Training Programs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser Visual Guidance group (Experimental): Will be tested using simulated laparoscopic tasks with the use of laser visual guidance
  Interventions: Device: Laser Visual Guidance
- Normal 2D vision group (Active Comparator): Will be tested using simulated laparoscopic tasks without the use of laser visual guidance
  Interventions: Device: 2 D vision

INTERVENTIONS:
Device: Laser Visual Guidance — Laparoscopic simulator training, tested with laser visual guidance
  Arms: Laser Visual Guidance group
Device: 2 D vision — Laparoscopic simulator training, tested without laser visual guidance
  Arms: Normal 2D vision group

SUMMARY:
"Laparoscopic simulation training with or without laser visual guidance -A randomised study" which investigates if the use of laser visual guidance can help the novices to learn the laparoscopic skills.

DETAILED DESCRIPTION:
Background: The loss of depth perception due to working in a three-dimensional space based on two-dimensional images is one of the challenging aspects of laparoscopy compared to conventional open surgery.

Objectives: To examine the effect of laser visual guidance on laparoscopic performance and cognitive load in a simulated setting for novices.

Methods: Randomised Clinical Trial- Laser visual guidance vs. normal 2 D vision.

Outcomes:

Primary outcome: Motor skills performance parameters-movement-time:

Cumulative instrument movement-time for both the right and left instrument for the test session,

Secondary outcome: 2) The overall composite score.

Exploratory outcomes: 3) The NASA Task Load index (NASA-TLX).

ELIGIBILITY:
Inclusion Criteria:

* Surgical novices / medical students enrolled at The Faculty of Health Science, University of Copenhagen.
* Participants are required to provide informed consent before inclusion.

Exclusion Criteria:

* Participation in prior studies involving laparoscopic training.
* Experience with laparoscopy surgery (having performed minimum one laparoscopic procedure as primary surgeon, including supervised procedures).
* No informed consent.
* Does not speak Danish on a conversational level.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Motor skills performance parameters (Cumulative Instrument movement-time) | 3 hours
  Cumulative Instrument movement-time

SECONDARY OUTCOMES:
The composite performance score (errors) | 3 hours
  points

OTHER OUTCOMES:
The NASA Task Load index (NASA-TLX). | 3 hours
  Work load index

CONTACTS AND LOCATIONS:
Overall Officials: Lars Konge, MD, PhD, Principal Investigator — Center for Clinical Education, Rigshospitalet,
Locations (1):
- Centre for Clinical Education, Copenhagen, Cooenhagen Ø, Denmark